CLINICAL TRIAL: NCT04821037
Title: Feasibility and Acceptability of a Virtual ACT-intervention in Nurses Working During the COVID-19 Pandemic (Pilot Study)
Brief Title: Nurse Health Pilot: Feasibility and Acceptability of a Virtual ACT-intervention in Nurses During COVID-19
Acronym: NHP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Prof. Dr. Andrew Gloster (Other)
Collaborators: State Secretariat for Education Research and Innovation, Switzerland (Other); ETH Zurich (Switzerland) (Other)
Responsible Party: Sponsor-Investigator, Prof. Dr. Andrew Gloster, Prof. Andrew Gloster, University of Basel
Organization: University of Basel (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: NHP
Record Dates: First submitted 2021-03-26; First posted 2021-03-29 (Actual); Last update posted 2021-06-02 (Actual); Status verified 2021-05

CONDITIONS: Stress
Keywords: stress; resilience; wellbeing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ACT (Experimental): A digitally-based ACT program will be conducted in two half-day workshops via meeting software (e.g. Zoom) consisting of:
  1. mindfulness exercises, for stress reduction and to guide nurses to observe their painful thoughts and feelings that they are attempting to avoid;
  2. ACT-metaphors, to let nurses realize the cost of struggling with psychological distress often create more distress;
  3. experiential exercises, to guide nurses to notice their own experiences in providing nursing care throughout their nursing career and explore any special qualities;
  4. explore the nurses' values with respect to different areas in their lives.
  Interventions: Behavioral: ACT

INTERVENTIONS:
Behavioral: ACT — Acceptance and Commitment Therapy

SUMMARY:
Frontline nurses increasingly face challenges between executing their jobs to the best of their ability and caring for their own physical and mental health. Such a stressful and fast-changing work environment impacts the nurses' psychological wellbeing, resulting in high levels of stress and burnout, which in turn negatively affects patient care and outcomes.

The aim of this study is to investigate whether a short virtual intervention, based on Acceptance and Commitment Therapy (ACT) and adapted to caregivers, can lead to a reduction in psychological distress that may be associated with caregiving during the COVID-19 pandemic.

The intervention will be held online in a group setting during two half-day workshops using a conference application (e.g. Zoom).

Note: This study is part of an international joint research project "Nurse Health" between the Faculty of Psychology (University of Basel) and the Nethersole School of Nursing (Chinese University of Hong Kong), funded by the Swiss State Secretariat for Education, Research and Innovation (SERI), with the Leading House for the Bilateral Science and Technology Cooperation Programme with Asia at ETH Zürich (Project No. COV_09_062020).

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years of age
* degree in nursing
* working 40% or higher in a team of nurses in the somatic area
* currently or previously in contact with COVID-19 patients
* working in Switzerland

Exclusion Criteria:

* working in non-somatic areas (e.g. psychiatry)
* working in non-hospital environments (e.g. home treatment)
* not owning an electronic device
* unable to understand and speak German

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2021-06-01 (Estimated); Primary Completion 2021-07-01 (Estimated); Study Completion 2021-08-01 (Estimated)

PRIMARY OUTCOMES:
Perceived Stress Scale (PSS-10) | 8 weeks
  Assessment of the perception of psychological stress (10 items)
General Anxiety Disorder Scale (GAD-7) | 8 weeks
  Assessment of the severity of anxiety (7 items)
Patient Health Questionnaire (PHQ-9) | 8 weeks
  Assessment of the severity of depression (9 items)
Maslach Burnout Inventory - Human Services Survey (MBI-HSS) | 8 weeks
  Assessment of the severity of burnout (22 items)
Mental Health Continuum Short Form (MHC-SF) | 8 weeks
  Assessment of perceived emotional wellbeing (14 items)
Psychological Flexibility Questionnaire (PsyFlex) | 8 weeks
  Assessment of psychological flexibility (6 items)
Valued Living Questionnaire (VLQ) | 8 weeks
  Assessment of the extent of valued living (10 items)
Mueller and McCloskey Satisfaction Scale (MMSS) | 8 weeks
  Assessment of nurses' job satisfaction (31 items)

SECONDARY OUTCOMES:
Program Attendance/ Attrition Rate | 8 weeks
  Percentage of program attendance
Homework Completion | 8 weeks
  Percentage of completed homework
Program Satisfaction | 8 weeks
  Rate of nurses' satisfaction with the program

CONTACTS AND LOCATIONS:
Overall Officials: Andrew T Gloster, Prof. Dr., Principal Investigator — Division of Clinical Psychology & Intervention Science, University of Basel
Locations (1):
- Faculty of Psychology, University of Basel, Basel, Canton of Basel-City, Switzerland

IPD SHARING:
Plan to Share IPD: No